CLINICAL TRIAL: NCT04222049
Title: Application of Vibration Wave Therapy to the Speech of Children Suffering From Cerebral Palsy and Dysarthria Using Neuro Transmission Cognitive Theory: Single Group Experimental Study
Brief Title: Application of Vibration Wave Therapy to the Children Suffering From Cerebral Palsy and Tongue Spastic Dysarthria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Science and Technology, Pakistan (Other)
Collaborators: Family Health Hospital Islamabad Pakistan (Unknown); Higher Education Commission (Pakistan) (Other)
Responsible Party: Principal Investigator, Aliya Ashraf Khan, principal investigator, National University of Science and Technology, Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUST-FHH-HEC
Record Dates: First submitted 2020-01-01; First posted 2020-01-09 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cerebral Palsy; Spastic Dysarthria
Keywords: Neurorehabilitation; Vibration; Neurotransmission; cerebral palsy; Dysarthria
MeSH Terms: conditions — Cerebral Palsy; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- spastic Tongue Dysarthria (Experimental): The purpose of gadget is to transmit the mechanical vibration waves to the brain of the subjects.
  Interventions: Device: Vibro Tactile Gadget

INTERVENTIONS:
Device: Vibro Tactile Gadget — The concept is to apply vibro tactile gadget to different nerve points which when applied transmit waves to the focused parts of brain which will result in blood flow and activation of dead cells. As a result some disabled part of the body because of those dead cells can show improvement.

SUMMARY:
Vibration therapy is the widely used in many neurological disorders for different type of problems. Recently, it is being used by researchers for the betterment of motor disorders and muscle movements of the cerebral palsy patients and significant results are obtained. Investigators are conducting this research to explore that whether this therapy can have some effect on the Spastic Tongue Dysarthria of the Cerebral Palsy patients.

DETAILED DESCRIPTION:
This study is going to be conducted in collaboration with Shahbaz Khalid Ranjha , Speech Language Pathologist, Family Health Hospital Islamabad who is the main person for the idea of the study and National University of Science & Technology. This study is funded by Higher Education Commission of Pakistan. Recruitment and Intervention Work will be carried out in Family Health Hospital. Special device is being designed for transmission of Vibration waves in Lab of the university. The device is capable to transmit vibration waves to the patient. Urdu language phonological and articulation test(TAAPU) will be used for assessment as it is specially designed for Urdu language population which will be the main focus. Investigators have defined speech parameters for analysis which will be collected before application of intervention, after 3 months and then at the end of the study. Parents assessment will be collected and noted through out the intervention.

ELIGIBILITY:
Inclusion Criteria:

* children having dysarthria due to cerebral Palsy
* Dysarthria due to damage in motor speech area/ broca area.
* Children having type Spastic Dysarthria

Exclusion Criteria:

Children diagnosed with following are excluded from our study

* Any speech disorders
* hearing impairments
* cleft palate
* tongue tie.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-06-14 (Actual)

PRIMARY OUTCOMES:
Child Historical Treatment Measurement | At Enrollment
  Socio demographic and Health related data is collected so that that efficacy of treatment under study can be calculated w.r.t pre treatment assessments
Change in phonological disorders using TAAPU Test for assessment of articulation and phonology in urdu language | At month 0, At month 03 and at month 06
  Scores for fronting, stopping, phonological disorders, final consonant deletion, Nasal assimilation and de-palatalization is calculated pre and post assessment through TAAPU(Test for assessment of articulation and phonology in urdu language).
Parent Assessment Checklist | At month 0
  A questionnaire is prepared for the child assessment by the parent.
Parent Assessment Checklist | At month 3
  A questionnaire is prepared for the child assessment by the parent.
Parent Assessment Checklist | At month 6
  A questionnaire is prepared for the child assessment by the parent.

SECONDARY OUTCOMES:
Parent Assessment Checklist | At month 01
  A questionnaire is prepared for the child assessment by the parent.
Parent Assessment Checklist | At month 02
  A questionnaire is prepared for the child assessment by the parent.
Parent Assessment Checklist | At month 04
  A questionnaire is prepared for the child assessment by the parent.
Parent Assessment Checklist | At month 05
  A questionnaire is prepared for the child assessment by the parent.
Change in phonological disorders using TAAPU Test for assessment of articulation and phonology in urdu language | At month 01 and At month 02
  Scores for fronting, stopping, phonological disorders, final consonant deletion, Nasal assimilation and de-palatalization is calculated pre and post assessment through TAAPU(Test for assessment of articulation and phonology in urdu language).

CONTACTS AND LOCATIONS:
Overall Officials: Shahbaz K Ranjha, MPhil, Study Director — Family Health Hospital Islamabad; Aliya A Khan, MS, Principal Investigator — National University of Science & Technology; Mohammad U Akram, Phd, Study Chair — National University of Science & Technology; Madeeha Nissar, MSc, Principal Investigator — Isra University Islamabad
Locations (1):
- Family Health Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
we will show the data to other researchers once study is completed and results are published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the publication of the results data will be available for researchers who can benefit from it whenever they want.
Access Criteria: Data will be shared to those researchers who want to continue research in the area